CLINICAL TRIAL: NCT01773148
Title: AXERA Access Safety and Efficacy Post Endovascular INtervention
Brief Title: Access Safety and Efficacy Post Endovascular Intervention
Acronym: ASPEN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Arstasis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC-03773
Record Dates: First submitted 2013-01-15; First posted 2013-01-23 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Cardiovascular Disease.
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arstasis Access System (AXERA) placement (Experimental): Placement of AXERA device in subjects undergoing common femoral artery access for PCI and/or PVI through a 5F or 6F introducer sheath.
  Interventions: Device: Arstasis Access System (AXERA)

INTERVENTIONS:
Device: Arstasis Access System (AXERA) — Placement of the AXERA device in the Femoral Artery.

SUMMARY:
The goal of this study is to assess the safety and effectiveness of the AXERA Access System in subjects undergoing Common Femoral Artery (CFA) access for Percutaneous Coronary Intervention (PCI) and/or Peripheral Vascular Intervention (PVI) through a 5 French (F) or 6F introducer sheath.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older.
* Subject is clinically indicated for a PCI or PVI involving access through a 5F or 6F introducer sheath in the femoral artery.
* Subject is able to ambulate without assistance prior to the procedure and can be expected to ambulate (20 feet) within 2 hours post procedure.
* Female subjects of child bearing potential must have a negative pregnancy test.

Exclusion Criteria:

* Subjects who are pregnant or lactating.
* Subject has a pre-existing severe non-cardiac systemic disease/illness or another reason that results in a projected life expectancy of less than 1 year.
* Subject has an active systemic or cutaneous infection or inflammation (e.g., septicemia at the time of the procedure).
* Subject has systemic hypertension unresponsive to treatment (>180mmHg systolic and >110mm diastolic).
* Subject has significant bleeding coagulopathy or platelet disorder, (INR> 2.0), including known thrombocytopenia (platelet count <100,000/µL), thrombasthenia, Von Willebrand's disease, Factor V deficiency, or anemia (hemoglobin <10 g/dL, or hematocrit <30%).
* Subject presents with chronic renal insufficiency (creatinine ≥3.0mg/dl).
* Subject presents with hemodynamic instability or is in need of emergent surgery or emergent procedure.
* Subject presents with ST elevation myocardial infarction.
* Subject presents with unstable angina or non-ST elevation myocardial infarction and has troponin level > 3 X upper limit of normal. There must be at least one troponin level drawn > 6 hours after onset of chest pain.
* Subject has received low molecular weight heparin < 8 hours before vascular access, glycoprotein IIb/IIIa inhibitor < 24 hours before vascular access, unfractionated heparin by infusion < 1 hour before vascular access, or parenteral heparin at anticoagulant dose (as opposed to DVT prophylaxis)< 6 hours before vascular access.
* Subjects who are clinically obese, defined as BMI >40.
* Subject has received femoral artery Vessel Closure Implant (VCI) (suture or staple) at the target access site.
* Subject has received femoral artery VCI (collagen/PEG/PGA) at the target access site within 90 days of AXERA procedure.
* Subject is unable to routinely walk at least 20 feet without assistance (e.g., requires a walker or wheelchair to mobilize, is leg amputee or has known paralysis) or unable to ambulate within 2 hours post procedure.
* Subject has had prior vascular surgery or vascular grafts at the target femoral artery access site.
* Subject has had a previous target femoral artery complication from angiography (such as pseudoaneurysm, Arteriovenous (AV) fistula, dissection), small CFA, abnormal, absent or weak distal ipsilateral pulse, or presenting with clinically significant peripheral vascular disease in the vicinity of the puncture.
* Subject has a high puncture (i.e. above the inferior reflection of the inferior epigastric artery).
* Subject has antegrade puncture.
* Subject has a stent in the ipsilateral common femoral artery.
* Subject is currently participating in an investigational drug or another device study that clinically interferes with the current study endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2012-12; Primary Completion 2015-03 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Events | Procedure through 30 day follow-up.
  Absence of major access site-related complications.
Device Success | Day 1-Day of Procedure.
  Defined as:
  * Successful placement of AXERA followed by procedural sheath
  * Achievement of hemostasis in conjunction with manual or mechanical compression

SECONDARY OUTCOMES:
Time to Hemostasis (TTH) | Immediately following procedural sheath removal.
  Elapsed time between sheath removal and first observed hemostasis.
Time to Ambulation (TTA) | Evaluated at any time after 2 hours post sheath removal, until the subject successfully ambulated.
  Elapsed time between sheath removal to time when subject stands and walks at least 20 feet without re-bleeding.
Time to Discharge, eligibility (TTD/e) | Evaluated following sheath removal and ambulation and physical examination of the access site demonstrating stable access site.
  Elapsed time between sheath removal and the time when subject is medically able to be discharged.
Time to Discharge, actual (TTD/a) | Evaluated following procedural sheath removal until actual discharge.
  Elapsed time between sheath removal and the actual time when subject is discharged.
Minor Adverse Events | Procedure through 30 day follow-up.
  Combined rate of minor vascular access-site related complications.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Dorogy, MD, Principal Investigator — The Medical Center of Central Georgia
Locations (17):
- United States (17):
  - Heart Center Research, LLC, Huntsville, Alabama
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Scripps Green, La Jolla, California
  - Loma Linda University Health, Loma Linda, California
  - Mercy Heart and Vascular Institute, Sacramento, California
  - St. Joseph's Medical Center, Stockton, California
  - Christiana Care, Newark, Delaware
  - Medical Center of Central Georgia, Macon, Georgia
  - Opelousas General Health System, Opelousas, Louisiana
  - Sinai Hospital, Baltimore, Maryland
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Northern Mississippi Medical Center, Tupelo, Mississippi
  - St. Rose Dominican, Las Vegas, Nevada
  - St. John Medical Center, Tulsa, Oklahoma
  - AnMed Health, Anderson, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Franciscan Research Center, Tacoma, Washington